CLINICAL TRIAL: NCT05721274
Title: The Last Mile - Community Engagement and Conditional Incentives to Accelerate Polio Eradication in Conflict-affected Areas of Pakistan
Brief Title: Community Engagement and Conditional Incentives to Accelerate Polio
Acronym: GLIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr Jai Kumar Das, Assistant Professor and Assistant Director, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-7125-20666
Record Dates: First submitted 2023-01-12; First posted 2023-02-09 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Polio; Immunization; Infection; Incentives
Keywords: Community engagment; Theory of change
MeSH Terms: conditions — Poliomyelitis; Infections

STUDY DESIGN:
Intervention Model Description: The intervention is based on behaviour change theory
Masking Description: Project team will keep liaison with key stakeholders, committee members, polio workers/supervisors and other relevant persons. Influential community members will conduct awareness and motivation activities. The messages would address reasons for OPV and routine vaccine refusals in the community and will be disseminated via health promotion materials and support groups organized by committees.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The study will adopt a pretest/post-test quasi-experimental design. The approach of the proposed project is to implement a participatory community engagement and demand creation strategy with trust-building community mobilization and a conditional community-based incentive scheme to reduce the refusals to vaccination and improve polio immunization coverage in intervention UCs. Clusters will be formed on a population of 1500-2000 in each intervention UC. Committees would be formed with approximately 5-7 prominent members of the community.
  Intervention Non-cash, incentives would be given and decided with consensus by UC committees and aim to improve infrastructure linked to health including water and sanitation and toilets in the community.
  Interventions: Behavioral: Community mobilization and Conditional community incentives
- Control arm (No Intervention): This would be the standard of care

INTERVENTIONS:
Behavioral: Community mobilization and Conditional community incentives — Non-cash, incentives would be given to clusters which improve the polio vaccine coverage and reduce the refusals and these incentives would be decided with consensus by community and costs would be shared
  Arms: Intervention

SUMMARY:
Immunization is one of the most cost-effective and successful public health strategy in reducing the health, economic and societal burden of many infectious diseases. Pakistan and Afghanistan remain the only countries where polio is endemic, and Pakistan reports the most cases in the world. Although the rate is lower than in previous years, the situation remains alarming. This study objective is to decrease polio vaccine refusals and zero-dose vaccines by motivating behaviour change

DETAILED DESCRIPTION:
Study Design:The study will adopt a pretest/post-test quasi-experimental approach with two intervention UCs and two control UCs. For each target, intervention SHRUC, a separate, matched control SHRUC of comparable size and location will be identified for eventual pre-post comparison. Children under-five will be eligible for inclusion.

Intervention: The intervention package will include community mobilization and incentivization. Clusters will be formed on a population of 2000-2500 in each intervention UC, thus approximately ten clusters in each. Project will form or liaise with community groups or committees (male and female) in each cluster, which are already operational in many parts of the target UCs. However, to focus on reducing polio vaccine refusals, our program will adopt a unique incentivization approach, preceded by trust-building community mobilization. Clusters will be determined based on the existing micro plans of the PPEP. Microplans are a population-based set of components, at UC-level, used by the program for delivering polio vaccination efficiently. Baseline and end-line surveys will be conducted in the target and control UCs.

Study Site: The study will be conduucted in district Karachi, Sindh and other in district Bannu, KP.

Intervention UCs: Haji Mureed Goth Karchi and Mira-Khel KP COntrol UCs : Nazivmabad UC 49 Karachi and Khwajamad- Bannu)

The research team will engage with multiple village/mohalla committees in the intervention UCs to address and eliminate misconceptions about polio. One-to-one meetings and group sessions which will be led by the committee members, to provide messages on childhood immunization with project-specific IEC material, will be held in each targeted cluster. These platforms would be helpful to identify and counsel their underlying fears and socio-psychological factors about the vaccines, such as painful neonatal experiences, mishandling, doubts, fear of vaccine-related side effects, distrust, etc.

The community-based incentives will be conditional based on the decrease in vaccine refusal rates within stipulated time. Communities successful in achieving these targets will be rewarded incentives to improve their infrastructure, including sanitation and hygiene, and water resources.

ELIGIBILITY:
Inclusion Criteria:

• Household with at least one child 0-59 months of age

Exclusion Criteria:

• Thise not willing to participate in study

Ages: 1 Day to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 840 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Vaccine refusals | at 9 months
  Number of polio vaccine refusals in polio campaign
Fully Immunized Children | at 9 months
  This would be children who are fully vaccinated appropriate to the age
IPV coverage | at 9 months
  this would be injectable polio vaccine coverage in children below five years of age

CONTACTS AND LOCATIONS:
Locations (1):
- Jai Das, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Das JK, Khan A, Tabassum F, Padhani ZA, Habib A, Mirani M, Rahman AR, Khan ZA, Rizvi A, Ahmed I, Bhutta Z. The Last Mile-Community Engagement and Conditional Incentives to Accelerate Polio Eradication in Pakistan: Study Protocol for a Quasi-Experimental Trial. Methods Protoc. 2023 Sep 8;6(5):83. doi: 10.3390/mps6050083. PMID 37736966